CLINICAL TRIAL: NCT04444037
Title: Impact of Optical Coherence Tomography Imaging on Decision-making During Percutaneous Coronary Intervention in Patients Presented With Acute Coronary Syndromes
Brief Title: Impact of OCT Imaging on Decision Making During PCI in ACS Patients
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Collaborators: Wakayama Medical University (Other)
Responsible Party: Principal Investigator, Amir Khalifa Mahfouz Khalifa, Principle investigator, Cardiology department, Assiut University
Other Study IDs: OCT in ACS patients
Record Dates: First submitted 2020-06-20; First posted 2020-06-23 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Acute Coronary Syndrome
Keywords: OCT, stent implantation
MeSH Terms: conditions — Acute Coronary Syndrome; Ornithine Carbamoyltransferase Deficiency Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OCT-guided PCI: PCI procedure was done with intra-coronary imaging OCT.
  Interventions: Device: OCT-guided PCI
- Angiography-guided PCI: PCI procedure was done without any intra-coronary imaging assistance, guided by angiography alone

INTERVENTIONS:
Device: OCT-guided PCI — using optical coherence tomography imaging to help PCI procedure
  Groups: OCT-guided PCI

SUMMARY:
Optical coherence tomography (OCT) provides valuable information to guide percutaneous coronary intervention (PCI) in acute coronary syndrome (ACS) regarding lesion preparation, stent sizing, and stent optimization.

DETAILED DESCRIPTION:
OCT can be used in acute coronary syndrome (ACS). ACS has more complex culprit lesion morphologies and larger extent of coronary atherosclerosis compared with stable coronary artery disease. The detailed vascular information obtained by OCT may impact PCI in ACS, and which may improve acute results and late outcomes of PCI. Stent expansion immediately after PCI is a strong predictor of late outcomes of PCI, and it is associated with late clinical outcomes in many previous trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients presented with acute coronary syndrome.
* PCI was done to them with stent implantation.

Exclusion Criteria:

* Multivessel PCI at the index procedure.
* Patients with ACS due to graft failure post CABG.
* Patients treated with no stent implantation.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient either underwent PCI with angiography alone or OCT guided and is grouped accordingly
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Percent difference in lumen expansion in stent treated lesion | Immediately after the procedure
  Compare residual percent diameter stenosis, percent area stenosis, and acute lumen gain between the two groups.

SECONDARY OUTCOMES:
Clinical outcomes at 1 year follow up | During 1 year following the index procedure
  Cardiac death, MI, clinical-driven target-lesion revascularization (TLR), and stroke

CONTACTS AND LOCATIONS:
Overall Officials: Yehia T Kishk, MD, Study Chair — Assiut University; Hossam H Ali, MD, Study Chair — Assiut University; Ahmed Abdel-Galeel, MD, Study Chair — Assiut University; Takashi Akasaka, MD, PhD, Study Chair — Wakayama Medical University
Locations (1):
- Wakayama Medical University, Wakayama, Japan

IPD SHARING:
Plan to Share IPD: No
Nothing

REFERENCES:
- [Background] Wu S, Liu W, Guo Y, Zeng Y, Zhou Z, Zhao Y, Liu Y, Shi D, Wang Z, Ge H, Wang J, Jin P, Zhou Y. The impact of acute coronary syndrome on late drug-eluting stents restenosis: Insights from optical coherence tomography. Medicine (Baltimore). 2017 Dec;96(52):e9515. doi: 10.1097/MD.0000000000009515. PMID 29384957
- [Background] Kubo T, Shinke T, Okamura T, Hibi K, Nakazawa G, Morino Y, Shite J, Fusazaki T, Otake H, Kozuma K, Ioji T, Kaneda H, Serikawa T, Kataoka T, Okada H, Akasaka T; OPINION Investigators. Optical frequency domain imaging vs. intravascular ultrasound in percutaneous coronary intervention (OPINION trial): one-year angiographic and clinical results. Eur Heart J. 2017 Nov 7;38(42):3139-3147. doi: 10.1093/eurheartj/ehx351. PMID 29121226
- [Background] Khalifa AKM, Kubo T, Ino Y, Terada K, Emori H, Higashioka D, Katayama Y, Takahata M, Shimamura K, Shiono Y, Matsuo Y, Tanaka A, Hozumi T, Akasaka T. Optical Coherence Tomography Comparison of Percutaneous Coronary Intervention Among Plaque Rupture, Erosion, and Calcified Nodule in Acute Myocardial Infarction. Circ J. 2020 May 25;84(6):911-916. doi: 10.1253/circj.CJ-20-0014. Epub 2020 Apr 18. PMID 32307358
- [Background] Kubo T, Shinke T, Okamura T, Hibi K, Nakazawa G, Morino Y, Shite J, Ino Y, Kitabata H, Shimokawa T, Akasaka T. Comparison between Optical COherence tomography guidance and Angiography guidance in percutaneous coronary intervention (COCOA): Study protocol for a randomized controlled trial. J Cardiol. 2018 Aug;72(2):170-175. doi: 10.1016/j.jjcc.2018.01.005. Epub 2018 Mar 2. PMID 29486964
- [Background] Otake H, Kubo T, Shinke T, Hibi K, Tanaka S, Ishida M, Kataoka T, Takaya T, Iwasaki M, Sonoda S, Ioji T, Akasaka T. OPtical frequency domain imaging vs. INtravascular ultrasound in percutaneous coronary InterventiON in patients with Acute Coronary Syndrome: Study protocol for a randomized controlled trial. J Cardiol. 2020 Sep;76(3):317-321. doi: 10.1016/j.jjcc.2020.03.010. Epub 2020 Apr 24. PMID 32340781
- [Background] TIMI Study Group. The Thrombolysis in Myocardial Infarction (TIMI) trial. Phase I findings. N Engl J Med. 1985 Apr 4;312(14):932-6. doi: 10.1056/NEJM198504043121437. No abstract available. PMID 4038784
- [Background] Ali ZA, Maehara A, Genereux P, Shlofmitz RA, Fabbiocchi F, Nazif TM, Guagliumi G, Meraj PM, Alfonso F, Samady H, Akasaka T, Carlson EB, Leesar MA, Matsumura M, Ozan MO, Mintz GS, Ben-Yehuda O, Stone GW; ILUMIEN III: OPTIMIZE PCI Investigators. Optical coherence tomography compared with intravascular ultrasound and with angiography to guide coronary stent implantation (ILUMIEN III: OPTIMIZE PCI): a randomised controlled trial. Lancet. 2016 Nov 26;388(10060):2618-2628. doi: 10.1016/S0140-6736(16)31922-5. Epub 2016 Oct 30. PMID 27806900
- [Background] Meneveau N, Souteyrand G, Motreff P, Caussin C, Amabile N, Ohlmann P, Morel O, Lefrancois Y, Descotes-Genon V, Silvain J, Braik N, Chopard R, Chatot M, Ecarnot F, Tauzin H, Van Belle E, Belle L, Schiele F. Optical Coherence Tomography to Optimize Results of Percutaneous Coronary Intervention in Patients with Non-ST-Elevation Acute Coronary Syndrome: Results of the Multicenter, Randomized DOCTORS Study (Does Optical Coherence Tomography Optimize Results of Stenting). Circulation. 2016 Sep 27;134(13):906-17. doi: 10.1161/CIRCULATIONAHA.116.024393. Epub 2016 Aug 29. PMID 27573032